CLINICAL TRIAL: NCT04125290
Title: US Post-Marketing Retrospective Observational Safety Study of Moxetumomab Pasudotox-tdfk (LUMOXITI)(TM)
Brief Title: US Post-Marketing Safety Study of Moxetumomab Pasudotox-tdfk (LUMOXITI)
Acronym: PROXY
Status: Terminated | Type: Observational
Why Stopped: Study stopped due to lack of recruitment.
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D3143R00004
Record Dates: First submitted 2019-09-13; First posted 2019-10-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hairy Cell Leukemia
Keywords: capillary leak syndrome; hemolytic uremic syndrome; renal toxicity; infusion-related reaction; electrolyte abnormalities; HCL and all relevant indications where LUMOXITI will be prescribed
MeSH Terms: conditions — Leukemia, Hairy Cell; Capillary Leak Syndrome; Hemolytic-Uremic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
This study is being conducted to satisfy a post-marketing requirement (PMR) to provide evidence characterizing 1) the safety of moxetumomab pasudotox-tdfk in patients who are 65 years of age and older and/or 2) the safety of moxetumomab pasudotox-tdfk in patients who have moderate renal impairment defined as an estimated GFR of 30-59 ml/min

DETAILED DESCRIPTION:
The pivotal Phase 3 study (Study 1053) supported full approval of moxetumomab pasudotox-tdfk from the US Food and Drug Administration (FDA) for the treatment of adult patients with relapsed or refractory hairy cell leukemia (HCL) who received at least two prior systemic therapies, including treatment with a PNA, on 13 September 2018. Since HCL is a rare disease, clinical research has limited information concerning the safety of moxetumomab pasudotox-tdfk in elderly patient populations and patients with moderate renal impairment.This study is being conducted to satisfy a post-marketing requirement (PMR) to provide evidence characterizing the safety of moxetumomab in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent, if required
* Patient received at least 1 dose of moxetumomab pasudotox-tdfk and has completed or discontinued the treatment
* Patient has a medical record available from the start of first dose of moxetumomab pasudotox tdfk

AND at least 1 of the following:

* Patient is ≥65 years old at the time of starting initial treatment with moxetumomab pasudotox-tdfk OR
* Adult (≥18 years old) patient has moderate renal impairment, at the time of starting initial treatment with moxetumomab pasudotox-tdfk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be patients who are prescribed moxetumomab-pasudotox-tdfk who are ≥65 years old at the time of starting initial treatment with moxetumomab pasudotox-tdfk or are ≥18 years old with moderate renal impairment defined as an estimated GFR of 30-59 ml/min, at the time of starting initial treatment with moxetumomab pasudotox-tdfk. These two populations may not be mutually exclusive.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Incident proportion of capillary leak syndrome | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.
Incident proportion of hemolytic uremic syndrome | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.
Incident proportion of renal toxicity | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.
Incident proportion of infusion related reactions | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.
Incident proportion of electrolyte and biochemical abnormalities | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.
  Electrolyte and biochemical abnormalities are defined as laboratory measurements of interest that exceed local laboratory standards
Incident proportion of other medical events related to moxetumomab pasudotox-tdfk interruption or discontinuation | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.
Incident proportion of other serious medical events that are life-threatening, resulting in hospitalizations and/or death | From day 1 of moxetumomab pasudotox-tdfk initiation up to 30 days after last dose of moxetumomab pasudotox-tdfk.

CONTACTS AND LOCATIONS:
Overall Officials: Archna Hale, Study Director — AstraZeneca; Juan Cuevas, Principal Investigator — SSM Health DePaul Hospital; Travis Arculeta, Principal Investigator — Rocky Mountain Cancer Centers; Roser Calvo, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Research Site, Bridgeton, Missouri

REFERENCES:
- [Background] Bouroncle BA. Thirty-five years in the progress of hairy cell leukemia. Leuk Lymphoma. 1994;14 Suppl 1:1-12. PMID 7820038
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Kreitman 2018, Leukemia https://doi.org/10.1038/s41375-018-0210-1
- [Background] Kreitman RJ, Cheson BD. Malignancy: Current Clinical Practice: Treatment of Hairy Cell Leukemia at the Close of the 20th Century. Hematology. 1999;4(4):283-303. doi: 10.1080/10245332.1999.11746452. PMID 11399570
- [Background] Kroft SH, Tallman MS, Shaw JM, Thangavelu M, Peterson LC. Myelodysplasia following treatment of chronic lymphocytic leukemia (CLL) with 2-chlorodeoxyadenosine (2-CdA). Leukemia. 1997 Jan;11(1):170. doi: 10.1038/sj.leu.2400523. No abstract available. PMID 9001435
- [Background] Leleu X, Soumerai J, Roccaro A, Hatjiharissi E, Hunter ZR, Manning R, Ciccarelli BT, Sacco A, Ioakimidis L, Adamia S, Moreau AS, Patterson CJ, Ghobrial IM, Treon SP. Increased incidence of transformation and myelodysplasia/acute leukemia in patients with Waldenstrom macroglobulinemia treated with nucleoside analogs. J Clin Oncol. 2009 Jan 10;27(2):250-5. doi: 10.1200/JCO.2007.15.1530. Epub 2008 Dec 8. PMID 19064987
- [Background] Seymour JF, Kurzrock R, Freireich EJ, Estey EH. 2-chlorodeoxyadenosine induces durable remissions and prolonged suppression of CD4+ lymphocyte counts in patients with hairy cell leukemia. Blood. 1994 May 15;83(10):2906-11. PMID 7910051
- [Background] Seymour JF, Talpaz M, Kurzrock R. Response duration and recovery of CD4+ lymphocytes following deoxycoformycin in interferon-alpha-resistant hairy cell leukemia: 7-year follow-up. Leukemia. 1997 Jan;11(1):42-7. doi: 10.1038/sj.leu.2400513. PMID 9001417
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3143R00004&attachmentIdentifier=345bc15f-f08f-4914-ac4b-c0a67c6d7fb6&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=